CLINICAL TRIAL: NCT02726438
Title: A Phase 1, Open-Label Pharmacokinetic Study to Investigate Drug Penetration in the Bone After Repeated Oral Administration of Debio 1450 to Patients Undergoing Hip Replacement Surgery
Brief Title: Drug Penetration Into Bone After Repeated Oral Administration of Debio 1450 to Patients Undergoing Hip Replacement Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1450-108; 226488 (Other: CRO)
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Bone Diseases, Infectious
MeSH Terms: conditions — Bone Diseases, Infectious | interventions — afabicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Debio 1450 (Experimental): Participants will receive 3 oral administrations of Debio 1450 at a dose of 240 mg approximately 12 hours apart. The last dose should be given approximately 2, 4, 6 or 12 hours prior to surgery with 3 patients each to be dosed at each of these time points.
  If the surgery is delayed by more than 12 hours postdose, the patients could receive up to 2 additional administrations (approximately 12 hours apart) to ensure that the last dose is administered between 2 and 12 hours before the surgery.
  Interventions: Drug: Debio 1450
- Calibration (No Intervention): A single participant will not receive the study drug, providing data to be used as calibration.

INTERVENTIONS:
Drug: Debio 1450 — Debio 1450, 40 mg, powder for oral solution, for reconstitution in 5% dextrose in water.
  Arms: Debio 1450

SUMMARY:
Debio 1450 is being developed for the treatment of staph (staphylococcal) infections. How fast and completely an antibiotic penetrates into bone is used to determine how effective it might be to treat infections related to bones or joints. Since bone has fewer blood vessels than other tissue (for example lung tissue or the skin), drugs have a harder time getting into them. It is important to find out how much of the antibiotic can get into the bone to help patients with bone infections.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to comply with restrictions related to food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding);
  3. the analysis of results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Bone to plasma ratio for Debio 1452 (the Debio 1450 active moiety) | at pre-last dose (predose of the 3rd dose), at 0.5, 1, 2, 3, 5, 8, 12 hours post-last dose (Dose 3) and at the time of bone resection (surgery); only at the time of bone resection for the calibration participant
  Bone/bone marrow/soft tissue/synovial fluid samples will be collected during surgery; time of resection will be used to calculate the elapsed time after last dosing.

SECONDARY OUTCOMES:
Plasma ratios for Debio 1452 | at pre-last dose (predose of the 3rd dose), at 0.5, 1, 2, 3, 5, 8, 12 hours post-last dose (Dose 3) and at the time of bone resection (surgery); only at the time of bone resection for the calibration participant
  Categories: Bone marrow:plasma; soft tissue:plasma; synovial fluid:plasma
Area under the curve at steady state (AUCτ) of Debio 1452 | at pre-last dose (predose of the 3rd dose), at 0.5, 1, 2, 3, 5, 8, 12 hours post-last dose (Dose 3) and at the time of bone resection (surgery); only at the time of bone resection for the calibration participant
Maximum observed plasma concentration (Cmax) of Debio 1452 | at pre-last dose (predose of the 3rd dose), at 0.5, 1, 2, 3, 5, 8, 12 hours post-last dose (Dose 3) and at the time of bone resection (surgery); only at the time of bone resection for the calibration participant
Measured concentration at the end of a dosing interval at steady state (Ctrough) of Debio 1452 | at pre-last dose (predose of the 3rd dose), at 0.5, 1, 2, 3, 5, 8, 12 hours post-last dose (Dose 3) and at the time of bone resection (surgery); only at the time of bone resection for the calibration participant

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - eStudySite, La Mesa, California
  - Mercury St Medical Group, PLLC, Butte, Montana

REFERENCES:
- [Derived] Menetrey A, Janin A, Pullman J, Overcash JS, Haouala A, Leylavergne F, Turbe L, Wittke F, Nicolas-Metral V. Bone and Joint Tissue Penetration of the Staphylococcus-Selective Antibiotic Afabicin in Patients Undergoing Elective Hip Replacement Surgery. Antimicrob Agents Chemother. 2019 Feb 26;63(3):e01669-18. doi: 10.1128/AAC.01669-18. Print 2019 Mar. PMID 30559136